CLINICAL TRIAL: NCT06169696
Title: Visual Interface System for Improved Navigation and Accessibility Through EEG, Allowing for an EEG-driven Mobility Platform Offering Wheelchair-enabled Engagement and Rehabilitation (EMPOWER): An Early Feasibility Study (EFS) of Safety and Efficacy in Subjects With Severe Quadriplegia
Brief Title: EMPOWER Early Feasibility Study: Non-invasive BCI to Control a Wheelchair for People With Paralysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Synaptrix Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SYNL-01-01
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Neurologic Disorder; Paralysis; Paralysis; Stroke; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries; Cervical Spinal Cord Injury; Tetraplegic; Paralysis; Quadriplegia/Tetraplegia
Keywords: Amyotrophic Lateral Sclerosis; Quadriplegia/Tetraplegia
MeSH Terms: conditions — Nervous System Diseases; Paralysis; Stroke; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries; Quadriplegia | interventions — Methods; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Group / Arm (Other): Use of non-invasive EEG headband device
  Interventions: Device: Intervention/Treatment

INTERVENTIONS:
Device: Intervention/Treatment — Non-invasive EEG headband device
  Other Names: Neuralis by Synaptrix Labs

SUMMARY:
Neuralis is an innovative assistive technology designed for individuals with severe neuromuscular conditions, enabling wheelchair control through EEG signals. This study aims to assess the safety, feasibility, and efficacy of Neuralis in restoring mobility and independence.

The device is a discreet EEG headset which specializes in decoding signals from visual cortex, allowing users to initiate precise wheelchair movements through focused attention. This research seeks to demonstrate Neuralis' potential in revolutionizing assistive technology by offering a non-invasive, user-friendly solution for individuals facing motor impairments, ultimately enhancing their quality of life.

DETAILED DESCRIPTION:
Neuralis, developed by Synaptrix Labs, is an innovative assistive technology engineered to restore mobility and independence for individuals grappling with severe neuromuscular conditions. This cutting-edge device operates through a discreet and non-invasive EEG headset, comprising strategically placed dry sensors at on the occipital lobe, precisely targeting the visual cortex region.

The key breakthrough lies in Neuralis' capability to extract brain activity from subtle eye movements. Through this interaction, Neuralis decodes subtle EEG signals, effectively translating them into precise wheelchair navigation commands.

The device interfaces seamlessly with a user-friendly Neuralis mobile app, serving as the central control hub. This intuitive application handles calibration settings, connectivity, and destination selections through a simplified visual click-based protocol. The slim BCI headset captures EEG data, transmitting it via Bluetooth to the connected smartphone. Subsequently, the data is relayed to a secure cloud server, which houses an advanced computational infrastructure employing edge computing principles for optimal response times.

Within this cloud environment, a proprietary machine learning pipeline for EEG decoding and intent classification operates. Certain latency-sensitive steps run on the phone, while the cloud handles additional model training and personalization, leveraging scalable processing power. This dynamic architecture ensures a swift and near-instantaneous translation of the user's movement intentions into seamless wheelchair maneuverability.

What sets Neuralis apart is its ability to deliver robust functionality in a discreet, user-friendly manner. Its lightweight construction, comprising only four sensors, maximizes comfort while capturing essential visual cortex signals vital for nimble maneuvering. This fusion of advanced neurotechnology and user-centric design positions Neuralis as a significant leap forward in assistive devices, bridging the gap between usability and high-performance functionality for individuals with severe neuromuscular conditions.

Neuralis is completely non-invasive and built from stable, off the shelf parts. All data is encrypted.

ELIGIBILITY:
Inclusion Criteria:

1. Severe quadriparesis
2. Able to give consent
3. Appropriate candidate for device
4. Able and willing to access all clinical testing and not impeded by geographical location
5. Proficient in English
6. Have a study partner

Exclusion Criteria:

1. History of seizures
2. History of epilepsy
3. Psychiatric or psychological disorder
4. No study partner or caregiver
5. Unable to provide evidence of COVID vaccination

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Device safety and efficacy | 1 month
  Number of patients who can comfortable and safely use device

CONTACTS AND LOCATIONS:
Locations (1):
- Synaptrix Labs, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers